CLINICAL TRIAL: NCT00151918
Title: A Multi-Centre, Open Label, Randomized, Parallel Group Pilot Study to Assess the Efficacy and Safety of Lanthanum Carbonate and Sevelamer Hydrochloride in Patients Receiving Haemodialysis for End Stage Renal Disease
Brief Title: Efficacy and Safety of Lanthanum Carbonate and Sevelamer Hydrochloride in Patients Receiving Haemodialysis for End Stage Renal Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD405-310; 2004-001608-11 (EudraCT Number)
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — lanthanum carbonate

INTERVENTIONS:
Drug: Lanthanum carbonate

SUMMARY:
The purpose of this study is to assess phosphate reduction and control in patients with End Stage Renal Disease treated with either lanthanum carbonate or sevelamer hydrochloride

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving haemodialysis for ESRD
* Patients must have received haemodialysis for chronic renal failure three times per week for at least the previous 2 months

Exclusion Criteria:

* Pregnant or lactating women
* Patients with clinically significant uncontrolled concurrent illness, a life-threatening malignancy or current multiple myeloma
* Patients who are HIV+
* Patients with any significant bowel obstruction, active inflammatory bowel disease, GI motility disorders, or a history of major GI surgery within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2005-01-07 (Actual); Primary Completion 2005-08-22 (Actual); Study Completion 2005-08-22 (Actual)

PRIMARY OUTCOMES:
Mean pre-dialysis serum phosphate level | The last 4 weeks of the treatment period (Weeks 5, 6, 7, & 8)

SECONDARY OUTCOMES:
Mean pre-dialysis serum calcium product | The last 4 weeks of the treatment period (Weeks 5, 6, 7, & 8)
Mean pre-dialysis calcium-phosphate product | The last 4 weeks of the treatment period (Weeks 5, 6, 7, & 8)
Average daily pill burden | Daily throughout for the 8 week Evaluation for Dose Adjustment Period up to the End of Study/ Withdrawal Visit.
Treatment emergent adverse events | Throughout the study period of approximately 7.5 months.
  Treatment-emergent adverse events (TEAEs) were defined as AEs that had an onset date and time on or after the date and time of the first dose of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda